CLINICAL TRIAL: NCT06618716
Title: Individual Differences in the Acute Response to Experimentally Induced Inflammation: Microcirculatory Changes and Psychological Predictors
Brief Title: Individual Differences in Acute Response to Experimental Inflammation: Microcirculatory Changes and Psychological Predictors
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Karolinska Institutet (Other); Stockholm University (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, Associate Professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2023-07974-01
Record Dates: First submitted 2024-09-12; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Inflammation Biomarkers; Inflammation
Keywords: Microcirculatory status; Sickness behaviour; Lipopolysaccharide; Non-invasive monitoring
MeSH Terms: conditions — Inflammation | interventions — endotoxin, Escherichia coli; Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endotoxin (Active Comparator): The USP (United States Pharmacopeia Convention) Endotoxin RS (LPS; Endotoxin Reference Standard, Escherichia coli, Pharmacopeia, Rockville, MD, US) will be ordered.and comes as a lyophilized (freeze-dried) powder, and each vial contains 10,000 USP Endotoxin Units. Each vial contains approximately 1 microgram of Endotoxin. The lyophilized LPS will be dissolved in 5mL sterile water to obtain a solution at 200 ng/mL. This solution will be aliquoted in 400μL (thus containing 80ng endotoxin) and stored at -20°C. Aliquots will be sent for microbial safety testing routine and verification of endotoxin concentration to a certified laboratory. On the study day, 2100μL of physiological saline (sterile, pyrogen-free isotonic NaCl solution) will be added to the aliquot to obtain a final concentration of 32 ng/mL. The amount of solution to inject will then be calculated according to the participant's weight [in mL = (0.8 x weight) / 32].
  Interventions: Biological: endotoxin escherichia coli (E. coli) lipopolysaccharide (LPS)
- Placebo (Placebo Comparator): An equivolume of sterile physiological saline (NaCl 0.9%) will be used as placebo.
  Interventions: Other: Placcebo

INTERVENTIONS:
Biological: endotoxin escherichia coli (E. coli) lipopolysaccharide (LPS) — Intravenous administration of endotoxin (0.8 ng/kg body weight)
  Arms: Endotoxin
Other: Placcebo — Placebo injection of 0.9% NaCl
  Arms: Placebo

SUMMARY:
The physiological and behavioral responses to inflammatory vary greatly between individuals. The knowlegde about what causes these differences is sparse but plausible explanations are variations in sensitivity to peripheral inflammation. The goal of the study is to understand microcirculatory changes in skin and their possible correlation with conventional measurements of sickness and disease in humans. A better understanding of possible psychological predictors of sickness behaviour is also warranted as it may affect the results.

The general aim of the study is to assess microcirculatory changes in skin of the face, chest, hands and feet using different optical imaging techniques, and to identify psychological predictors in the acute behavioral response to experimentally induced inflammation. The participants are healthy volunteers in the age of 18-40 years of both sex/genders. The main questions to answer are:

1. How do acute inflammation change microcirculation in the skin as measured by temperature, red blood cell concentration, blood flow and spectral changes correlated with fluids and other proteins.
2. Can a stronger behavioral response to experimental endotoxemia be predicted by psychological factors of the individuals?

It is a blinded with-in subject, crossover design where the participants will receive placebo-injection with saline on one study day and LPS-injection the other study day in a randomized order.

Participants will on the study days

* Fill in psychometric questionnaires
* Be measured with bio-optical imaging methods at regular intervalls.
* Be monitored with regular medical parameters such as blood pressure, oxygen saturation, puls etc When the volunteers feel recovered and the medical staff are confident of the recovery the volunteers will be discharged.

DETAILED DESCRIPTION:
Background Acute illness manifest itself not only by physiological responses such as e.g. fever, pain and nausea, but is often accompanied by psychological and behavioral changes such as sleep/wake disturbances, fatigue, loss of appetite and depression. The physiological and behavioral responses to inflammatory activation vary greatly between individuals. The knowledge about what causes these differences is sparse, but plausible explanations are variations in sensitivity to peripheral inflammation and inflammation-induced brain changes. As the skin is readily accessible, it provides an appropriate site to assess microvascular reactivity during inflammation. Moreover, recent technological advances have provided simple and non-invasive methods to assess skin microvascular function. Therefore, human cutaneous circulation could be used as a surrogate marker of systemic microvascular function in inflammation. In the present study, we use experimentally induced immunological activation in healthy humans to study microcirculatory skin changes as well as behavioral predictors of individual sensitivity to an acute inflammatory stimulus.

The model of experimental endotoxemia to induce acute inflammation The model of experimental endotoxemia is a well-accepted and frequently used model to study the neuropsychiatric effects of pro-inflammatory cytokines, both in animals and in humans. The model is based on the sterile activation of the immune system, obtained by intravenous injection of an endotoxin, lipopolysaccharide (LPS), a wall component of gram-negative bacteria such as E. coli. Injection of LPS will affect the functionality of the vascular endothelium. Positioned at the interface between circulating blood and surrounding tissue, endothelial cells, which line the inner walls of blood vessels, play a crucial role in the response to pathogens. The endothelium serves various functions essential for maintaining organ homeostasis, including vasoregulation, selective vascular permeability, and providing an anticoagulant surface. However, during infection, the normal physiological functions of the endothelium are disrupted, contributing to the organ failure characteristic of sepsis. Importantly, the response to inflammation during experimental endotoxemia differs substantially across individuals. This holds for the degree of increase in inflammatory cytokines, the neural response, as well as the behavioral changes that entail inflammation. It should be noted that the neuropsychiatric response to inflammation is not explained fully by the magnitude of the inflammatory response, indicating that other factors are involved. Recent research points toward the importance of top-down mechanisms in modifying the effect of inflammation on behavior. Such mechanisms might include pre-existent emotional status and beliefs about the intensity of which one will become sick after an infection. Identifying the predictors of a heightened behavioral response to inflammation would help identifying markers of inflammation-associated neuropsychiatric vulnerability, but this has rarely been investigated.

General aim The general aim of the study is to assess microcirculatory changes in skin of the face, chest, hands and feet using different optical imaging techniques, and to identify psychological predictors in the acute behavioral response to experimentally induced inflammation.

Primary research questions

The main research questions are:

1. to assess how acute inflammation affects:

   * the microcirculation in skin such as face, chest, arms, hands and feet as investigated with different non-invasive optical imaging techniques:
   * Core temperature changes
   * Facial temperature changes
   * Changes in equivalents to red blood cell concentration and blood flow
   * Spectral changes in skin possibly correlated with fluids and other proteins affected by microcirculatory changes
2. to assess whether a stronger behavioral response (i.e. sickness behavior, negative mood, fatigue, anxiety, pain) to experimental endotoxemia is predicted by:

   * higher interoceptive sensitivity as measured by self-report and an objective task (heartrate discrimination task);
   * less cognitive resilience (i.e. self-efficacy, optimism, perseverance, coping strategies, ability to update beliefs in the fact of contradictory evidence);
   * worse baseline emotional status (i.e. trait anxiety, fatigue, perceived stress);
   * stronger health anxiety and disgust tendencies;
   * Sociocultural factors that have been found to relate to sickness behavior, such as stoic endurance of pain and discomfort, familism, individualism, and collectivism;
   * baseline biological motion pattern (walking speed, rigidity of gait, and slumped posture);

Methods Research principals The research principals are Region Östergötland, Karolinska Institutet and Stockholm University, Sweden. Data collection will be conducted at the Emergency Medicine Research Center (EMRC). Processing of data will be conducted at EMRC, Region Östergötland, Karolinska Institutet and Stockholm University.

Study design The study will be conducted at the Emergency Medicine Research Center at the University Hospital of Linköping. The study will follow a double-blind within-subject crossover placebo-controlled design. All subjects will receive an intravenous administration of LPS at a dose of up to 0.8 ng/kg body weight once, and an intravenous administration of placebo once, in a randomized order and with at least 4 weeks of wash-out period. Upon arrival, volunteers will be placed on a hospital bed in a single room and a catheter will be placed in the forearm or hand to avoid multiple needle insertion. A urine sample for pregnancy testing and drug screening will be obtained for safety reasons. The participants will then complete the baseline questionnaires, and the baseline blood sample will be drawn. After the baseline assessments, volunteers will receive the LPS or placebo injection. Vital signs (pulse, blood pressure, blood-oxygen saturation, respiratory frequency) will be continuously monitored and recorded at 30-minute intervals. Body temperature will be monitored and recorded every 30 minutes with regular tympanic thermometer, as well as continuously, using bio-optical imaging techniques. Blood samples will be taken approximately every hour to measure the inflammatory response (see "assessments - inflammatory markers from blood samples" below). Bio-optical imaging will be performed once before injection and at several occasions after the injection. Web-based questionnaires will be completed regularly to measure the sickness and emotional response will be completed by the participants just after acquisition of blood samples. Several behavioral tasks will be conducted during the study day. Volunteers will be discharged 6-10 hrs or when considered recovered by medical staff, after the injection, following a medical examination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 18-40 years-old
* Consent form signed
* Having a Swedish personal identification number (personnummer)

Exclusion Criteria:

* Non-fluent in Swedish
* Unable to read
* Unable or unwilling to provide informed consent
* BMI below 18.5 or above 25 kg/m2
* Smoking
* Excessive alcohol consumption
* Pregnancy or breastfeeding
* Positive on drug screening
* Current somatic disease including skin disease affecting the measurement areas
* Current depression, anxiety, sleep disturbances or other psychiatric illnesses
* Abnormal blood analyses: abnormal clinical levels in blood cell counts, hemoglobin, sodium, potassium, chloride, calcium, phosphate, creatinine, blood urea nitrogen, uric acid, glucose, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transpeptidase, bilirubin, thromboplastin time and partial thromboplastin time
* High-sensitivity C-reactive protein > 10 mg/L.
* History of cardiovascular, pneumological, immune disease
* Moderate viral or bacterial infection in the past two weeks
* Severe and/or long-term COVID-19: positive SARS-CoV-2 PCR-test or antigen-test and/or history of symptoms since February 2020 indicative of infection with SARS-CoV-2 (fever, cough, sore throat, runny or blocked nose, nausea, muscle pain, shortness of breath), which was of high intensity and/or of long duration (≥ 8 weeks).
* Recent vaccination (within previous two weeks)
* Abnormal cardiovascular measurements
* Current or previous cancer
* Any concomitant medication other than contraceptives (14 days prior to the start and throughout the study period)
* Shift work or irregular sleep-wake cycle (within 14 days of the study period)
* Needle anxiety or blood phobia
* Invisible veins in the antecubital area of the arms or very difficult blood sampling (self-reported or experienced during screening).
* Previous participation in a study involving administration of LPS

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
How does inflammation affect the behavioral response? | Baseline
  Behavioral response in psychometric tests measuring sickness behavior, negative mood, anxiety and fatigue on Likert scales.
How does inflammation affect the behavioral response? | during the intervention
  Behavioral response in psychometric tests measuring sickness behavior, negative mood, anxiety and fatigue on Likert scales.
How does inflammation affect the behavioral response? | after the intervention
  Behavioral response in psychometric tests measuring sickness behavior, negative mood, anxiety and fatigue on Likert scales.
Microcirculatory changes in skin measured with bio-optical instruments | Baseline
  - Red Blood Cell tissue fraction - %
Microcirculatory changes in skin measured with bio-optical instruments | during the intervention
  - Red Blood Cell tissue fraction - %
Microcirculatory changes in skin measured with bio-optical instruments | after the intervention
  - Red Blood Cell tissue fraction - %
Microcirculatory changes in skin measured with bio-optical instruments | Baseline
  - Blood flow - mm/s
Microcirculatory changes in skin measured with bio-optical instruments | during the intervention
  Blood flow - mm/s
Microcirculatory changes in skin measured with bio-optical instruments | after the intervention
  - Blood flow - mm/s
Changes in skin and core temperature | Baseline
  Measured in degrees Celsius
Changes in skin and core temperature | during the intervention
  Measured in degrees Celsius
Changes in skin and core temperature | after the intervention
  Measured in degrees Celsius

CONTACTS AND LOCATIONS:
Overall Officials: Rani Toll, PhD, Principal Investigator — Department of Emergency Medicine in Linköping, and Department of Biomedical and Clinical Sciences, Linköping University, Linköping, Sweden
Locations (1):
- Department of emergency medicine, Linköping University Hospital, Region Östergötland, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Pseudomized data on the psychometric tests and kinetic tests will be shared with other researchers.
Supporting Information: Study Protocol, CSR
Time Frame: 17/9/24 to 31/12/29
Access Criteria: The co-investigators from Karolinska Institutet Stockholm University will be able to access IPD and supporting information.